CLINICAL TRIAL: NCT01547117
Title: Dietary Salt in Postural Tachycardia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alfredo Gamboa, Research Associate Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 111261; R01HL102387 (NIH)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-01

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: POTS; Orthostatic Intolerance; Orthostatic Tachycardia
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance | interventions — Blood Volume; Carbon Monoxide; Erythrocyte Count

STUDY DESIGN:
Intervention Model Description: Randomization tables will be used to determine whether the 10 mEq sodium/day or 300 mEq sodium/day diet will be consumed first. Both diets will be completed on each subject (randomized crossover study), so all of the study procedures (after screening) will be repeated.
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Sodium Level (Experimental): POTS and healthy controls will be randomly assigned the order of dietary sodium levels. All procedures are performed at both levels. The high sodium diet will provide 300 milliequivalents (mEq) sodium/day.
  Interventions: Radiation: Blood Volume; Radiation: Total Blood Volume; Procedure: Exercise Capacity Test - Bicycle; Procedure: Posture Study
- Low Sodium Dietary Level (Experimental): POTS and healthy controls will be randomly assigned the order of dietary sodium levels. All procedures are performed at both levels. The low sodium diet will provide 10 mEq sodium/day.
  Interventions: Radiation: Blood Volume; Radiation: Total Blood Volume; Procedure: Exercise Capacity Test - Bicycle; Procedure: Posture Study

INTERVENTIONS:
Radiation: Blood Volume — we will measure the amount of hemoglobin and myoglobin in the body by a procedure called CO rebreathing. One teaspoon of blood is taken before and after a small amount of CO has been absorbed into the bloodstream.
  Other Names: carbon monoxide (CO)-red blood cell (RBC) Blood Volume
Radiation: Total Blood Volume — Using injection of iodinated I-131 tagged human serum albumin nominally 25 microcuries of radiation, blood samples are drawn before and 30 minutes after injection.
  Other Names: DAXOR
Procedure: Exercise Capacity Test - Bicycle — subjects breath room air through a mouthpiece and exhale the air into a tube that connects to a machine (metabolic cart) that analyzes carbon dioxide and oxygen content, which allows the investigator to calculate the amount of oxygen they are using under resting and exercise conditions.
  Other Names: VO2 Max (maximal oxygen consumption)
Procedure: Posture Study — Blood pressure and heart rate will be measured while supine and then while standing for up to 30 minutes. Blood will be drawn in each position to measure hormones that regulate blood pressure and blood volume.
  Other Names: Standing Orthostatic Challenge

SUMMARY:
Patients with POTS may not adequately expand their plasma volume in response to a high-sodium (Na+) diet. Mechanisms involved in the regulation of plasma volume, such as the renin-angiotensin-aldosterone system and renal dopamine, may be impaired in POTS and may respond inappropriately to changes in dietary sodium.The purpose of this study is to determine (1) whether a high dietary sodium level appropriately expands plasma volume in POTS; (2) whether plasma renin activity and aldosterone are modified appropriately by changes in dietary sodium in POTS; and (3) whether patients with POTS have improvements in their orthostatic tachycardia and symptoms as a result of a high dietary sodium level.

DETAILED DESCRIPTION:
Study Day 1

* Start 150 milliequivalents (mEq) Na+/day diet (POTS patients as inpatients; healthy control subjects with clinical research center (CRC)- provided outpatient diet)
* Start a 24h urine collection (for Na+, K+, Cr, fractionated catecholamines)
* Blood work
* Blood volume - carbon monoxide rebreathing

Study Day 2

* Complete 24h urine
* Start STUDY DIET (10 mEq Na+/day or 300 mEq Na+/day in a random order) after 3 meals of 150 mEq Na+/day are complete; water ad lib

Study Day 3 - 5

* Continue STUDY DIET; water ad lib
* On Day 5, a 24 hr holter combined ECG monitor will be placed on the subjects.

Study Day 6

* Continue STUDY DIET; water ad lib
* Remove 24h Holter combined ECG monitor and BP monitor from subject
* Start a 24h urine collection (for Na+, K+, Cr, fractionated catecholamines)
* Complete questionnaires
* Nothing by mouth (NPO) after midnight for study next day

Study Day 7 (BIG DAY)

* Awaken early (~6am) to void (still collecting 24h urine)
* Patient returns to bed, IV catheter inserted
* Posture Study (in morning; between 7-8am ideally)
* Blood pressure and heart rate will be measured while supine and then while standing for up to 30 minutes
* We will draw 3 tablespoons of blood in each body position to measure hormones that regulate blood pressure and blood volume
* Hormones to verify the subject's phase of menstrual cycle
* Serum/plasma aliquots for future analysis
* Subjects will rate symptoms during supine period and at end of stand using Vanderbilt Orthostatic Symptoms Score (VOSS)
* Total Blood Volume (DAXOR)- using injection of iodinated I-131 tagged human serum albumin nominally 25 micro-Ci of radiation blood samples drawn through IV catheter before injection and for ~30 minutes post-injection (total - 25 ml)
* This will be done after supine assessment, but before standing the subject up
* Autonomic Function Test with Cardiac Output and Brief Tilt
* The subject will be tilted up to 60-75 degrees head-up tilt for up to 10 minutes to measure the changes in heart rate and blood pressure and symptoms with upright challenge.
* Blood volume - carbon monoxide rebreathing
* Exercise Capacity Test (in the afternoon) Will estimate maximal oxygen consumption (VO2 max) This test will be conducted on a stationary bicycle. Effort will be gradually increase while expired air is measured during exhaustive physical work.

All procedures are repeated at least a month later with the 2nd level of dietary salt. (Randomized to high or low salt to the first phase, the second phase is the remaining level)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with postural tachycardia syndrome by the Vanderbilt Autonomic Dysfunction Center
* Increase in heart rate ≥30 beats/min with position change from supine to standing (10 minutes)
* Chronic symptoms consistent with POTS that are worse when upright and get better with recumbence
* Age between 18-50 years old
* Non-smokers
* Premenopausal patients with POTS and healthy volunteers
* Only female participants are eligible.
* Since 80-90% of POTS patients are female, and there can be differences in measures with the menstrual cycle, including a small number of males might introduce a significant amount of noise.
* Able and willing to provide informed consent

Exclusion Criteria:

* Smokers
* Overt cause for postural tachycardia, i.e., acute dehydration
* Significant cardiovascular, pulmonary, hepatic, or hematological disease by history or screening results
* Pregnant (positive pregnancy test) or breastfeeding
* Hypertension defined as supine resting BP>145/95 mmHg off medications or needing antihypertensive medication
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies or an unpredictable schedule
* Unable to give informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-03; Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo J Gamboa, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Laurin JKH, Oyewunmi OA, Garland EM, Gamboa A, Nwazue VC, Paranjape SY, Black BK, Okamoto LE, Shibao CA, Biaggioni I, Robertson D, Diedrich A, Dupont WD, Sheldon RS, Raj SR. Adrenal gland response to adrenocorticotropic hormone is intact in patients with postural orthostatic tachycardia syndrome. Auton Neurosci. 2023 Sep;248:103105. doi: 10.1016/j.autneu.2023.103105. Epub 2023 Jun 24. PMID 37393658
- [Derived] Garland EM, Gamboa A, Nwazue VC, Celedonio JE, Paranjape SY, Black BK, Okamoto LE, Shibao CA, Biaggioni I, Robertson D, Diedrich A, Dupont WD, Raj SR. Effect of High Dietary Sodium Intake in Patients With Postural Tachycardia Syndrome. J Am Coll Cardiol. 2021 May 4;77(17):2174-2184. doi: 10.1016/j.jacc.2021.03.005. PMID 33926653

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy Participants: 17 were enrolled and randomized. 1 withdrew due to scheduling. 1 withdrew with migraines in phase 1 (low Na+). 2 withdrew in phase 1 (high Na+): 1 unable to tolerate study diet and another had difficulty cooperating with investigators.
  Postural Tachycardia Syndrome (POTS): 21 were enrolled and randomized. 6 withdrew before baseline due to age (1), pregnancy (1), prohibited meds (3), and scheduling (1). A 7th patient withdrew during phase 1 (high Na+) due to family illness.
Groups:
- Healthy Participants-Low Na+ Then High Na+: Healthy controls were randomly assigned the order of dietary sodium (Na+) levels. After baseline labs on Day 0 and 1 day on diet with 150 milliequivalents (mEq) sodium/day, 12 participants consumed low Na+ diet (10 mEq sodium/day; LS) for 6 days followed in at least 1 month by baseline labs, 1 day of 150 mEq sodium/day and 6 days of high Na+ diet (300 mEq sodium/day; HS). All procedures were performed at both levels.
- Healthy Participants-High Na+ Then Low Na+: Healthy controls were randomly assigned the order of dietary sodium (Na+) levels. After baseline labs on Day 0 and 1 day on diet with 150 mEq sodium/day, 5 participants consumed high Na+ diet (300 mEq sodium/day; HS) for 6 days followed in at least 1 month by baseline labs, 1 day of 150 mEq sodium/day and 6 days of low Na+ diet (10 mEq sodium/day; LS). All procedures were performed at both levels.
- Patients With POTS-Low Na+ Then High Na+: Patients with POTS were randomly assigned the order of dietary sodium (Na+) levels. After baseline labs on Day 0 and 1 day on diet with 150 mEq sodium/day, 10 participants consumed low Na+ diet (10 mEq sodium/day; LS) for 6 days followed in at least 1 month by baseline labs, 1 day of 150 mEq sodium/day and 6 days of high Na+ diet (300 mEq sodium/day; HS). All procedures were performed at both levels.
- Patients With POTS-High Na+ Then Low Na+: Patients with POTS were randomly assigned the order of dietary sodium (Na+) levels. After baseline labs on Day 0 and 1 day on diet with 150 mEq sodium/day, 11 participants consumed high Na+ diet (300 mEq sodium/day; HS) for 6 days followed in at least 1 month by baseline labs, 1 day of 150 mEq sodium/day and 6 days of low Na+ diet (10 mEq sodium/day; LS). All procedures were performed at both levels.
Period: Overall Study
Arm/Group | Healthy Participants-Low Na+ Then High Na+ | Healthy Participants-High Na+ Then Low Na+ | Patients With POTS-Low Na+ Then High Na+ | Patients With POTS-High Na+ Then Low Na+
Started | 12 | 5 | 10 | 11
Phase 1 Baseline Labs | 12 | 4 (1 healthy control was unable to find time to schedule study) | 8 (2 patients with POTS did not discontinue medication that was prohibited by protocol.) | 7 (1 patient with POTS did not discontinue medication that was prohibited by protocol, 1 patient was unable to find time to schedule the study, 1 was noted to be too old to participate, and 1 became pregnant between enrollment and the start of phase 1.)
Phase 1-150 mEq Sodium/Day | 12 | 4 | 8 | 7
Phase 1-start Low Sodium or High Sodium Diet | 12 | 4 | 8 | 7
Phase 1-finish | 11 (1 healthy control withdrew with migraines during phase 1 (low Na+).) | 2 (2 healthy controls withdrew during phase 1 (high Na+): 1 unable to tolerate study diet and another with difficulty cooperating with investigators..) | 8 | 6 (1 patient with POTS withdrew during phase 1 due to a family illness.)
Phase 2-150 mEq Sodium/Day | 11 | 2 | 8 | 6
Phase 2-start Low Sodium or High Sodium Diet | 11 | 2 | 8 | 6
Phase 2-finish | 11 | 2 | 8 | 6
Completed | 11 | 2 | 8 | 6
Not Completed | 1 | 3 | 2 | 5
Not completed — Physician Decision | 0 | 1 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: 14 patients with Postural Tachycardia Syndrome (POTS) and 13 Controls underwent testing while on a High Sodium Diet and while on a Low Sodium Diet, administered in a randomly assigned order. Baseline data were collected prior to starting the first dietary phase.
Groups:
- Healthy Participants-Low Na+ Then High Na+: Healthy controls were randomly assigned the order of dietary sodium (Na+) levels. After 1 day on diet with 150 mEq sodium/day, participants consumed low Na+ diet (10 mEq sodium/day; LS) for 6 days followed in at least 1 month by 1 day of 150 mEq sodium/day and 6 days of high Na+ diet (300 mEq sodium/day; HS). All procedures were performed at both levels.
- Healthy Participants-High Na+ Then Low Na+: Healthy controls were randomly assigned the order of dietary sodium (Na+) levels. After 1 day on diet with 150 mEq sodium/day, participants consumed high Na+ diet (300 mEq sodium/day; HS) for 6 days followed in at least 1 month by 1 day of 150 mEq sodium/day and 6 days of low Na+ diet (10 mEq sodium/day; LS). All procedures were performed at both levels.
- Patients With POTS-Low Na+ Then High Na+: Patients with POTS were randomly assigned the order of dietary sodium (Na+) levels. After 1 day on diet with 150 mEq sodium/day, participants consumed low Na+ diet (10 mEq sodium/day; LS) for 6 days followed in at least 1 month by 1 day of 150 mEq sodium/day and 6 days of high Na+ diet (300 mEq sodium/day; HS). All procedures were performed at both levels.
- Patients With POTS-High Na+ Then Low Na+: Patients with POTS were randomly assigned the order of dietary sodium (Na+) levels. After 1 day on diet with 150 mEq sodium/day, participants consumed high Na+ diet (300 mEq sodium/day; HS) for 6 days followed in at least 1 month by 1 day of 150 mEq sodium/day and 6 days of low Na+ diet (10 mEq sodium/day; LS). All procedures were performed at both levels.
- Total: Total of all reporting groups
Arm/Group | Healthy Participants-Low Na+ Then High Na+ | Healthy Participants-High Na+ Then Low Na+ | Patients With POTS-Low Na+ Then High Na+ | Patients With POTS-High Na+ Then Low Na+ | Total
Number analyzed (Participants) | 11 | 2 | 8 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6) | 35 (10) | 36 (9) | 32 (6) | 33 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 8 | 6 | 27
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 10 | 2 | 8 | 5 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 9 | 2 | 8 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 2 | 8 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Plasma Volume
Description: Plasma volume (PV) was determined by the indicator tracer-dilution technique, using the DAXOR Blood Volume Analyzer (BVA)-100 system (DAXOR Corporation), on Day 7 of the low sodium and high sodium dietary interventions. Outcome data are the absolute values for PV on Day 7 for each diet.
Time Frame: after 7 days of each dietary sodium level
Population: No data analysis for 1 healthy control who had poor venous access on Day 7 of the high sodium diet.
Measure: Median (Inter-Quartile Range); unit: mL
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Plasma Volume: Using injection of iodinated I-131 tagged human serum albumin, blood samples were drawn before and 30 minutes after injection on Day 7 of the diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Plasma Volume: Using injection of iodinated I-131 tagged human serum albumin, blood samples were drawn before and 30 minutes after injection on Day 7 of the diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the low sodium diet.
  Plasma Volume: Using injection of I-131 tagged human serum albumin, blood samples were drawn before and 30 minutes after injection on Day 7 of the diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the high sodium diet.
  Plasma Volume: Using injection of I-131 tagged human serum albumin, blood samples were drawn before and 30 minutes after injection on Day 7 of the diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.
Number analyzed (Participants) | 13 | 12 | 14 | 14
mL | 2805 [2445 to 2949] | 3032 [2620 to 3482] | 2362 [2161 to 2715] | 2633 [2468 to 2961]

2. Secondary Outcome: Magnitude of Suppression of Plasma Renin Activity (From Low Sodium to High Sodium Diets)
Description: Whether upright plasma renin activity was modified appropriately by changes in dietary sodium in POTS & healthy controls. Outcome data are the absolute values for upright plasma renin activity on Day 7 of each diet.
Time Frame: Upright blood samples were collected after up to 30 minutes of standing on the 7th day of each dietary sodium intervention
Population: Healthy Controls on Low Sodium diet - 1 missing blood sample; Healthy Controls on High Sodium diet - 3 missing blood samples, 2 samples with insufficient volume for analysis; POTS patients on Low Sodium diet - 1 missing blood sample; POTS patients on High Sodium diet - 2 missing blood samples
Measure: Median (Inter-Quartile Range); unit: ng/mL/hr
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Upright plasma renin activity was measured in blood samples collected after up to 30 minutes of standing on the 7th day of low sodium diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Upright plasma renin activity was measured in blood samples collected after up to 30 minutes of standing on the 7th day of high sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the low sodium diet.
  Upright plasma renin activity was measured in blood samples collected after up to 30 minutes of standing on the 7th day of low sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the high sodium diet.
  Upright plasma renin activity was measured in blood samples collected after up to 30 minutes of standing on the 7th day of high sodium diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.
Number analyzed (Participants) | 12 | 8 | 13 | 12
ng/mL/hr | 7.8 [3.3 to 13.9] | 1.0 [.8 to 1.9] | 24.4 [10.1 to 26.7] | 2.7 [.7 to 4.8]

3. Other Pre Specified Outcome: Magnitude of Suppression of Serum Aldosterone (From Low Sodium to High Sodium Diets)
Description: Whether upright serum aldosterone was modified appropriately by changes in dietary sodium in POTS patients & healthy controls. Outcome data are the absolute values for upright serum aldosterone on Day 7 of each diet.
Time Frame: as for outcome 2
Population: Samples were analyzed from each participant
Measure: Median (Inter-Quartile Range); unit: ng/dL
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Upright serum aldosterone was measured in blood samples collected after up to 30 minutes of standing on the 7th day of low sodium diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Upright serum aldosterone was measured in blood samples collected after up to 30 minutes of standing on the 7th day of high sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the low sodium diet.
  Upright serum aldosterone was measured in blood samples collected after up to 30 minutes of standing on the 7th day of low sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the high sodium diet.
  Upright serum aldosterone was measured in blood samples collected after up to 30 minutes of standing on the 7th day of high sodium diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.
Number analyzed (Participants) | 13 | 13 | 14 | 14
ng/dL | 444 [277 to 515] | 74 [52 to 129] | 455 [359 to 650] | 64 [52 to 91]

4. Other Pre Specified Outcome: Magnitude of Orthostatic Tachycardia
Description: Whether the magnitude of the heart rate increase that occurs in patients with POTS when moving from a supine to an upright position is attenuated by a High Sodium diet relative to a Low Sodium diet.
  Heart rate was assessed after overnight rest and fasting after midnight, following at least 60 minutes of lying quietly. Heart rate was then measured at intervals after subjects had been standing for up to 30 minutes (as tolerated). Orthostatic tachycardia was calculated as the difference between standing and lying heart rates. Data are presented for 5 minutes standing (or maximal stand if <5 minutes) since several patients were unable to stand for 10 minutes.
  Data in POTS patients were compared to that of Healthy Controls.
Time Frame: Supine and upright heart rates were measured on Day 7 of High Sodium and Low Sodium diet.
Population: Data is not included for 1 patient with POTS on a Low Sodium diet since that patient was unable to stand for even 1 minute.
Measure: Median (Inter-Quartile Range); unit: beats per minute
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Supine and upright heart rate were measured on the 7th day of low sodium diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Supine and upright heart rate were measured on the 7th day of high sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the low sodium diet.
  Supine and upright heart rate were measured on the 7th day of low sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the high sodium diet.
  Supine and upright heart rate were measured on the 7th day of high sodium diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.
Number analyzed (Participants) | 13 | 13 | 13 | 14
beats per minute | 23 [19 to 36] | 19 [11 to 32] | 60 [55 to 64] | 46 [32 to 55]

5. Other Pre Specified Outcome: Upright Symptom Score
Description: Whether upright symptoms were improved in patients with POTS on a High Sodium diet relative to a Low Sodium diet.
  Patients were asked to report their standing symptom burden at the end of the Stand portion of the posture study, using the Vanderbilt Orthostatic Symptoms Scale (VOSS). They rated the severity of nine symptoms (palpitations, lightheadedness, mental confusion, blurred vision, shortness of breath, tremulousness, chest discomfort, headache, and nausea) on a scale from a minimum of 0 (reflecting an absence of symptoms) to a maximum of 10. The sum of the scores for the 9 symptoms was used to measure orthostatic symptom burden. Higher scores represent worse symptoms.
Time Frame: Upright symptoms were assessed on the 7th day of diet.
Population: Upright symptom scores were inadvertently not obtained for the following number of participants:
  Healthy Participants on Low Sodium diet: 3 Healthy Participants on High Sodium diet: 2 Patients with POTS on Low Sodium diet: 5 Patients with POTS on High Sodium diet: 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Upright symptoms were assessed on the 7th day of low sodium diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Upright symptoms were assessed on the 7th day of high sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the low sodium diet.
  Upright symptoms were assessed on the 7th day of low sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the high sodium diet.
  Upright symptoms were assessed on the 7th day of high sodium diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.
Number analyzed (Participants) | 10 | 11 | 9 | 8
score on a scale | 1 [0 to 4] | 0 [0 to 3] | 30 [18 to 39] | 19 [10 to 26]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through discharge on the last day of phase 2 of the study. This would have been Day 8 if Low Sodium diet or Day 7 if High Sodium diet.
Description: Adverse event information was collected for any untoward or unfavorable medical occurence in a participant including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Events were self-reported by participants.
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the low sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.: Patients were randomly assigned the order of dietary sodium levels. Results below were after the high sodium diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 1/13 | 0/14 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B (N=13) | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B (N=13) | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. (N=14) | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet. (N=14)
mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 — Participant notified the PI that a mass had been discovered on her pineal gland during a brain MRI for another research study. We do not believe that the mass is related to any study procedures undertaken as part of this research protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT01547117/Prot_SAP_000.pdf